**Official study title:** Does Focusing on Body Functionality Improve Body Image Among Women Who Have Undergone Bariatric Surgery?

Study title for participants: Positief Lichaamsbeeld (Positive Body Image)

Ethics approval number: ERCPN-167\_03\_05\_2016 (approved June 2nd, 2016)

**Document:** Informed consent sheet

## **Declaration of Consent**

For participation in the study entitled,

"Positief Lichaamsbeeld"
[Positive Body Image]

I have been informed about this study. I have read the written information. I have had the opportunity to ask questions about this study. I have had the opportunity to think about my participation in this study, and my participation is entirely voluntary. I have the right to withdraw my consent and to terminate my participation in this study, without needing to provide a reason.

| I agree to take part in this study: | |
|---|---|
| Name: | |
| Birth date: | |
| Signature: | Date: |
| The responsible researcher (see below) declares that the participant named above has been fully informed of this study. | |
| Name: | |
| Role: | |
| Signature: | Date: |